CLINICAL TRIAL: NCT02561221
Title: Promoting Successful Weight Loss in Primary Care in Louisiana
Acronym: PROPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana State University Health Sciences Center Shreveport (Other); Tulane University (Other); Ochsner Health System (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Xavier University of Louisiana. (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director for Population and Public Health Sciences, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2015-052; PCORI#OB-1402-10977 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: primary care; pragmatic trial; weight loss; overweight; diet; physical activity; PCORI
MeSH Terms: conditions — Obesity; Weight Loss; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Counseling (Experimental): Patients in the Lifestyle Counseling Arm attended weekly (16 in-person) sessions in the first six months, followed by monthly sessions for the remaining 18 months. The behavioral intervention was delivered by a trained health coach embedded in the primary care clinic. Primary Care Practitioners in the experimental arm received a series of webinars on obesity science to help them manage and treat patients with obesity.
  Interventions: Behavioral: Lifestyle Counseling
- Usual Care (No Intervention): Patients assigned to the usual care arm continued to interact with their Primary Care Practitioners according to their usual schedule, and received a series of newsletters on topics of interest, including importance of sleep for health, brain and memory health, goal setting, smoking cessation, etc. Primary Care Practitioners in the usual care arm received a webinar describing the current Centers for Medicare and Medicaid (CMS) approach to reimbursing for obesity treatment, and a reminder informational brochure was sent to the Primary Care Practitioners each year.

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Trained health coaches delivered the active intervention - a comprehensive, "high-intensity" program, as recommended first-line therapy by the 2013 American Heart Association/American College of Cardiology/The Obesity Society Guidelines.
  Arms: Lifestyle Counseling

SUMMARY:
The primary aim of this trial is to develop and test the effectiveness of a 24 month, patient-centered, pragmatic and scalable obesity treatment program delivered within primary care, inclusive of an underserved population. Half of the clinics received a behavioral intervention delivered in a primary care setting and half of the clinics received usual care.

DETAILED DESCRIPTION:
This study is a cluster-randomized, two-arm controlled trial in primary care settings. A total of 18 primary care clinics inclusive of low income populations with a high percentage of African Americans from urban and rural areas across Louisiana were randomized to either 1) intervention or 2) usual care. The sample includes 803 patients with obesity (BMI 30-50 kg/m2) (18 clinics, median of 40.5 patients / clinic). The primary aim of this trial is to develop and test the effectiveness of a 24 month, patient-centered, pragmatic and scalable obesity treatment program delivered within primary care, inclusive of an underserved population. Patients in the intervention arm attended weekly (16 in-person) sessions in the first six months, followed by monthly sessions for the remaining 18 months. The behavioral intervention was delivered by a trained health coach embedded in the primary care clinic. Primary Care Practitioners in the intervention arm received a series of webinars on obesity science to help them manage and treat obese patients. Patients assigned to the usual care arm will continue to interact with their Primary Care Practitioner according to their usual schedule, and will receive a series of newsletters on topics of interest, including importance of sleep for health, brain and memory health, goal setting, smoking cessation, etc. Primary Care Practitioners in the usual care arm received a webinar describing the current Centers for Medicare and Medicaid Services (CMS) approach to reimbursing for obesity treatment, and a reminder informational brochure will be sent to the Primary Care Practitioners each year. Patients in both arms were assessed on primary and secondary outcome measures at baseline, and at 6, 12, 18 and 24 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20.0 - 75.0 years
* BMI 30.0 - 50.0 kg/m2
* Able to provide written informed consent
* Willing to change diet, physical activity and weight
* Patient of a participating clinic
* Able to participate in scheduled sessions

Exclusion Criteria:

* Currently participating in a weight loss program
* Current use of weight loss medication or recent weight loss (>10 lbs in last 6 months)
* Plans to move from the area within 2 years
* Given birth within the past year, is currently pregnant or plans to become pregnant within 2 years
* Past bariatric surgery or plans for bariatric surgery within 2 years
* Current major depression
* History of suicidal behavior or diagnosed eating disorder (bulimia, anorexia)
* Hospitalization for mental disorder or substance abuse in the previous year
* Active cancer (except prostate, skin and thyroid if approved by physician)
* Serious arrhythmias or cardiomyopathy
* Severe congestive heart failure
* Stroke or heart attack in previous six months
* Chronic Inflammatory conditions, including but not limited to severe arthritis, lupus, or inflammatory bowel disease(i.e. Crohn's disease or ulcerative colitis)
* Disease that is life threatening or that can interfere with or be aggravated by exercise or weight loss
* Discretion of primary care physician or principal investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2016-04; Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request and upon approval of the PROPEL Publications Committee. Data will be made available 1 year after publication of the primary outcomes manuscript. A data sharing statement and the protocol are available at: https://www.nejm.org/doi/full/10.1056/NEJMoa2007448
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon reasonable request to the Principal Investigator 1 year after the publication of the Primary Outcomes manuscript.
Access Criteria: Access to the data must be approved by the PROPEL Publications Committee.

REFERENCES:
- [Result] Katzmarzyk PT, Martin CK, Newton RL Jr, Apolzan JW, Arnold CL, Davis TC, Denstel KD, Mire EF, Thethi TK, Brantley PJ, Johnson WD, Fonseca V, Gugel J, Kennedy KB, Lavie CJ, Price-Haywood EG, Sarpong DF, Springgate B. Promoting Successful Weight Loss in Primary Care in Louisiana (PROPEL): Rationale, design and baseline characteristics. Contemp Clin Trials. 2018 Apr;67:1-10. doi: 10.1016/j.cct.2018.02.002. Epub 2018 Feb 8. PMID 29408562
- [Result] Myers CA, Martin CK, Newton RL Jr, Apolzan JW, Arnold CL, Davis TC, Price-Haywood EG, Katzmarzyk PT. Cardiovascular Health, Adiposity, and Food Insecurity in an Underserved Population. Nutrients. 2019 Jun 19;11(6):1376. doi: 10.3390/nu11061376. PMID 31248113
- [Result] Katzmarzyk PT, Martin CK, Newton RL Jr, Apolzan JW, Arnold CL, Davis TC, Price-Haywood EG, Denstel KD, Mire EF, Thethi TK, Brantley PJ, Johnson WD, Fonseca V, Gugel J, Kennedy KB, Lavie CJ, Sarpong DF, Springgate B. Weight Loss in Underserved Patients - A Cluster-Randomized Trial. N Engl J Med. 2020 Sep 3;383(10):909-918. doi: 10.1056/NEJMoa2007448. PMID 32877581
- [Result] Hochsmann C, Dorling JL, Martin CK, Newton RL Jr, Apolzan JW, Myers CA, Denstel KD, Mire EF, Johnson WD, Zhang D, Arnold CL, Davis TC, Fonseca V, Lavie CJ, Price-Haywood EG, Katzmarzyk PT; PROPEL Research Group. Effects of a 2-Year Primary Care Lifestyle Intervention on Cardiometabolic Risk Factors: A Cluster-Randomized Trial. Circulation. 2021 Mar 23;143(12):1202-1214. doi: 10.1161/CIRCULATIONAHA.120.051328. Epub 2021 Feb 9. PMID 33557578
- [Result] Dorling JL, Martin CK, Yu Q, Cao W, Hochsmann C, Apolzan JW, Newton RL, Denstel KD, Mire EF, Katzmarzyk PT. Mediators of weight change in underserved patients with obesity: exploratory analyses from the Promoting Successful Weight Loss in Primary Care in Louisiana (PROPEL) cluster-randomized trial. Am J Clin Nutr. 2022 Oct 6;116(4):1112-1122. doi: 10.1093/ajcn/nqac179. PMID 35762659
- [Result] Katzmarzyk PT, Mire EF, Martin CK, Newton RL Jr, Apolzan JW, Price-Haywood EG, Denstel KD, Horswell R, Chu ST, Johnson WD; PROPEL Research Group. Comparison of weight loss data collected by research technicians versus electronic medical records: the PROPEL trial. Int J Obes (Lond). 2022 Aug;46(8):1456-1462. doi: 10.1038/s41366-022-01129-9. Epub 2022 May 6. PMID 35523955
- [Result] Katzmarzyk PT, Denstel KD, Martin CK, Newton RL Jr, Apolzan JW, Mire EF, Horswell R, Johnson WD, Brown AW, Zhang D; PROPEL Research Group. Intraclass correlation coefficients for weight loss cluster randomized trials in primary care: The PROPEL trial. Clin Obes. 2022 Aug;12(4):e12524. doi: 10.1111/cob.12524. Epub 2022 Apr 12. PMID 35412010
- [Result] Katzmarzyk PT, Apolzan JW, Gajewski B, Johnson WD, Martin CK, Newton RL Jr, Perri MG, VanWormer JJ, Befort CA. Weight loss in primary care: A pooled analysis of two pragmatic cluster-randomized trials. Obesity (Silver Spring). 2021 Dec;29(12):2044-2054. doi: 10.1002/oby.23292. Epub 2021 Oct 29. PMID 34714976
- [Result] Katzmarzyk PT, Mire EF, Martin CK, Newton RL, Apolzan JW, Denstel KD, Johnson WD; PROPEL Research Group. Physical activity and weight loss in a pragmatic weight loss trial. Int J Obes (Lond). 2023 Mar;47(3):244-248. doi: 10.1038/s41366-023-01260-1. Epub 2023 Jan 26. PMID 36702913
- [Derived] Katzmarzyk PT, Mire EF, Horswell R, Chu ST, Zhang D, Martin CK, Newton RL, Apolzan JW, Price-Haywood EG, Fort D, Carton TW, Denstel KD; PROPEL Research Group. Four-year follow-up of weight loss maintenance using electronic medical record data: The PROPEL trial. Obes Sci Pract. 2024 Oct 19;10(5):e70017. doi: 10.1002/osp4.70017. eCollection 2024 Oct. PMID 39429541
- [Derived] Hochsmann C, Martin CK, Apolzan JW, Dorling JL, Newton RL Jr, Denstel KD, Mire EF, Johnson WD, Zhang D, Arnold CL, Davis TC, Fonseca V, Thethi TK, Lavie CJ, Springgate B, Katzmarzyk PT; PROPEL Research Group. Initial weight loss and early intervention adherence predict long-term weight loss during the Promoting Successful Weight Loss in Primary Care in Louisiana lifestyle intervention. Obesity (Silver Spring). 2023 Sep;31(9):2272-2282. doi: 10.1002/oby.23854. Epub 2023 Aug 8. PMID 37551762
- [Derived] Apolzan JW, Martin CK, Newton RL Jr, Myers CA, Arnold CL, Davis TC, Johnson WD, Zhang D, Hochsmann C, Fonseca VA, Denstel KD, Mire EF, Springgate BF, Lavie CJ, Katzmarzyk PT; PROPEL Research Group. Dietary intake during a pragmatic cluster-randomized weight loss trial in an underserved population in primary care. Nutr J. 2023 Aug 2;22(1):38. doi: 10.1186/s12937-023-00864-7. PMID 37528391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen primary care clinics were randomized equally to either the Intensive Lifestyle Intervention or Usual Care. Patients received the intervention to which their clinic was assigned. Study enrollment occurred from April 2016 to September 2017. Patients completed a pre-screener and attended a screening visit which included the consent process and measurement to determine height and weight for BMI among other eligibility criteria. Patients were enrolled upon baseline visit completion.
Units Other Than Participants: Primary care clinics
Period: Overall Study
Arm/Group | Lifestyle Counseling | Usual Care
Started | 452; 9 Primary care clinics | 351; 9 Primary care clinics
Month 6 | 386; 9 Primary care clinics | 340; 9 Primary care clinics
Month 12 | 365; 9 Primary care clinics | 326; 9 Primary care clinics
Month 18 | 357; 9 Primary care clinics | 316; 9 Primary care clinics
Completed | 362; 9 Primary care clinics | 308; 9 Primary care clinics
Not Completed | 90; 0 Primary care clinics | 43; 0 Primary care clinics

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Patients assigned to the usual care arm continued to interact with their Primary Care Practitioners according to their usual health care schedule, and received a series of newsletters on topics of interest, including importance of sleep for health, brain and memory health, goal setting, smoking cessation, etc.
  Primary Care Practitioners in the usual care arm received a webinar describing the current Centers for Medicare and Medicaid (CMS) approach to reimbursing for obesity treatment, and a reminder informational brochure was sent to the Primary Care Practitioners each year.
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Usual Care | Total
Number analyzed (Participants) | 452 | 351 | 803
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.7) | 50.1 (13.6) | 49.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398 | 280 | 678
  Male | 54 | 71 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 332 | 208 | 540
  White | 95 | 113 | 208
  Other | 25 | 30 | 55
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.3 (4.6) | 37.2 (4.8) | 37.2 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (Percent Change)
Description: Body weight is measured in light indoor clothes.
Time Frame: Percent (%) Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Lifestyle Counseling: Patients in the Intensive Lifestyle Intervention Arm attended weekly (16 in-person) sessions in the first six months, followed by monthly sessions for the remaining 18 months. The behavioral intervention was delivered by a trained health coach embedded in the primary care clinic. Primary Care Practitioners in the experimental arm received a series of webinars on obesity science to help them manage and treat patients with obesity.
  Intensive Lifestyle Intervention: Trained health coaches delivered the active intervention - a comprehensive, "high-intensity" program, as recommended first-line therapy by the 2013 American Heart Association/American College of Cardiology/The Obesity Society Guidelines.
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
percent change | -4.99 [-6.02 to -3.96] | -0.48 [-1.57 to 0.61]

2. Secondary Outcome: Waist Circumference
Description: Waist circumference is measured mid-way between the iliac crest and the lower rib margin.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
cm | -4.42 [-5.44 to -3.41] | 0.71 [-0.35 to 1.78]

3. Secondary Outcome: Systolic Blood Pressure
Description: Resting systolic blood pressures is measured.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mmHg | 1.94 [-0.75 to 4.63] | 0.41 [-2.43 to 3.26]

4. Secondary Outcome: Fasting Plasma Glucose
Description: Glucose is measured in the fasted state with a point-of-care device.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mg/dL | -1.25 [-5.65 to 3.15] | -0.33 [-4.61 to 3.94]

5. Secondary Outcome: Total Cholesterol
Description: Blood lipids/cholesterol are measured in the fasted state with a point-of-care device.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mg/dL | 4.64 [0.45 to 8.82] | -1.26 [-5.38 to 2.87]

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function
Description: The PROMIS-29 physical function sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a better outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A positive change score indicates improvement while a negative change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 0.82 [-0.16 to 1.79] | -0.39 [-1.39 to 0.62]

7. Secondary Outcome: PROMIS-29 Anxiety
Description: The PROMIS-29 Anxiety sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a worse outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | -0.92 [-2.29 to 0.46] | -0.53 [-1.95 to 0.89]

8. Secondary Outcome: PROMIS-29 Depression
Description: The PROMIS-29 Depression sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a worse outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | -0.18 [-1.17 to 0.81] | 0.64 [-0.34 to 1.63]

9. Secondary Outcome: PROMIS-29 Fatigue
Description: The PROMIS-29 Fatigue sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a worse outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | -2.82 [-4.06 to -1.59] | -1.03 [-2.28 to 0.22]

10. Secondary Outcome: PROMIS-29 Sleep Disturbance
Description: The PROMIS-29 sleep disturbance sub-scale includes 4 questions and scores ranges from 4 to 20 (higher values represent a worse outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | -1.25 [-2.45 to -0.05] | -0.35 [-1.59 to 0.89]

11. Secondary Outcome: PROMIS-29 Social Functioning
Description: The PROMIS-29 social roles sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a better outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A positive change score indicates improvement while a negative change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 1.57 [0.55 to 2.60] | 0.15 [-0.87 to 1.17]

12. Secondary Outcome: PROMIS-29 Pain Interference
Description: The PROMIS-29 pain interference sub-scale includes 4 questions and scores range from 4 to 20 (higher values represent a worse outcome). Transformed scores were used in analysis. Norm-based scores were calculated so that a score of 50 represents the mean or average of the reference population. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | -1.06 [-2.22 to 0.10] | 0.21 [-0.95 to 1.37]

13. Secondary Outcome: PROMIS-29 Pain Intensity
Description: The PROMIS-29 pain intensity sub-scale includes 1 question and scores range from 1 to 10 (higher values represent a worse outcome). A negative change score indicates improvement while a positive change score indicates worsening from baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
units on a scale | -0.02 [-0.35 to 0.30] | 0.21 [-0.12 to 0.53]

14. Secondary Outcome: Impact of Weight on Quality of Life-Lite (IWQOL-L) Total Score
Description: Impact of Weight on Quality of Life-Lite (IWQOL-L) measure consists of a total score and five subscales--physical function, self-esteem, sexual life, public distress, and work. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The total transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 11.02 [9.04 to 13.00] | 4.36 [2.34 to 6.39]

15. Secondary Outcome: IWQOL-L Physical Function
Description: The IWQOL-L physical function sub-scale includes 11 questions. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 12.31 [9.55 to 15.06] | 4.11 [1.24 to 6.97]

16. Secondary Outcome: IWQOL-L Self Esteem
Description: The IWQOL-L self-esteem sub-scale includes 7 questions. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 14.39 [11.66 to 17.12] | 7.62 [4.88 to 10.36]

17. Secondary Outcome: IWQOL-L Sexual Life
Description: The IWQOL-L sexual life sub-scale includes 4 questions. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 14.32 [11.00 to 17.65] | 4.49 [1.18 to 7.80]

18. Secondary Outcome: IWQOL-L Public Distress
Description: The IWQOL-L public distress sub-scale includes 5 questions. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 5.38 [2.86 to 7.89] | 2.41 [-0.20 to 5.02]

19. Secondary Outcome: IWQOL-L Work/Daily Activity
Description: The IWQOL-L work/daily activity sub-scale includes 4 questions. Transformed scores used in analyses were calculated so that scores are on a scale of 0 to 100. The transformed score ranges from 0 to 100 with higher change scores indicating greater improvement from Baseline.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
score on a scale | 5.48 [3.22 to 7.75] | 1.47 [-0.83 to 3.76]

20. Secondary Outcome: Body Weight (Absolute Change)
Description: Body weight is measured in light indoor clothes.
Time Frame: Absolute (kg) Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
kg | -5.43 [-6.52 to -4.34] | -0.91 [-2.07 to 0.24]

21. Secondary Outcome: Diastolic Blood Pressure
Description: Resting diastolic blood pressures is measured.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mmHg | -0.61 [-2.39 to 1.17] | -0.64 [-2.53 to 1.24]

22. Secondary Outcome: High-density Lipoprotein Cholesterol
Description: Blood lipids/cholesterol are measured in the fasted state with a point-of-care device.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mg/dL | 4.16 [2.78 to 5.54] | -0.44 [-1.81 to 0.94]

23. Secondary Outcome: Low-density Lipoprotein Cholesterol
Description: Blood lipids/cholesterol are measured in the fasted state with a point-of-care device.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mg/dL | 3.22 [-0.85 to 7.29] | -0.17 [-4.17 to 3.83]

24. Secondary Outcome: Triglycerides
Description: Blood lipids/cholesterol are measured in the fasted state with a point-of-care device.
Time Frame: Change from Baseline to Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 452 | 351
mg/dL | -11.23 [-22.02 to -0.44] | -5.58 [-16.39 to 5.23]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Lifestyle Counseling | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/452 | 1/351
Serious Adverse Events (participants affected / at risk) | 48/452 | 35/351
Other Adverse Events (participants affected / at risk) | 35/452 | 46/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Counseling (N=452) | Usual Care (N=351)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low White Blood Cell Count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach Ulcers (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vertigo/Dizziness (General disorders) | 0 (0) | 1 (1)
Severe Dehydration (General disorders) | 1 (1) | 1 (1)
Low Electrolytes/Minerals (General disorders) | 1 (1) | 0 (0)
Gallbladder Issues/Stones (Hepatobiliary disorders) | 1 (1) | 1 (1)
Otorhinolaryngological Infection (Infections and infestations) | 0 (0) | 1 (1)
Intestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory System Infection (Infections and infestations) | 3 (4) | 2 (2)
Allergic Reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Broken Bone (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mid- or Post-Surgical Complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Hyperglycemic Event (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycemic Event (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malignant Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Grand Mal Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Attempted Suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Enlarged Uterus (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hernia (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Penile Implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 5 (5) | 0 (0)
Musculoskeletal Surgery (Surgical and medical procedures) | 3 (3) | 2 (3)
Preventive Brain Bypass Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric Sleeve (Surgical and medical procedures) | 1 (1) | 0 (0)
Cyst Removal (Surgical and medical procedures) | 0 (0) | 2 (2)
Preventive Mastectomy and Reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Heller Myotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Occlusion (Vascular disorders) | 3 (3) | 1 (1)
Hypertensive Event (Vascular disorders) | 4 (5) | 1 (1)
Hypotensive Event (Vascular disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Counseling (N=452) | Usual Care (N=351)
Otorhinolaryngological Infection (Infections and infestations) | 20 (26) | 27 (35)
Respiratory System Infection (Infections and infestations) | 15 (19) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02561221/Prot_SAP_000.pdf